CLINICAL TRIAL: NCT03569566
Title: The Impact of Age, Genes, Training and History of Tickbourne Disease on Endurance Performance in Elite Endurance Athletes.
Brief Title: Performance Determinants Factors in Elite Endurance Athletes.
Status: Completed | Type: Observational
Sponsor: University of South-Eastern Norway (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/2522
Record Dates: First submitted 2018-05-28; First posted 2018-06-26 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2021-12

CONDITIONS: Exercise Physiology
Keywords: Age; Genes; Training volume; Training intensity; Tick-bourne disease; Endurance performance; Elite endurance athletes
MeSH Terms: interventions — Aging; Genes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples will be taken, and will be used for the following purposes:
  * DNA isolation and analysis: DNA genome will be isolated from white blood cells. This DNA genome will be contained in a biobank - Exercise Genetics. Well-known genetic variations in genes will be tested showing relevance to training adaptations (ACE, ACTN3 etc.). Only known polymorphisms will be investigated.
  * Exosome isolation from plasma: We will isolate exosomes from plasma by the ultracentrifugation method. We will investigate the volume and specific types of exosomes, in relation to the training intervention. We also want to examine the exosome-cargo, like miRNA, protein content, mRNA and DNA content.
  * Isolation of antibodies from plasma: We want to investigate antibodies to examine potential on-going disease, recently disease or earlier disease of Barbesia, Anaplasma or other actual tick-borne agens. We also want to isolate DNA from blood and use real-time PCR for anaplasma and Neo Ehrlichia analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elite endurance athletes: Cross-country skiers at high national level
  Interventions: Other: Age, Genes, Training, Tickbourne Disease and Endurance

INTERVENTIONS:
Other: Age, Genes, Training, Tickbourne Disease and Endurance — Testing of genes, exosomes, physiological variables, tick-bourne disease markers, observation of training modality and performance

SUMMARY:
Several studies have investigated determinant factors for endurance performance among different athletes, untrained individuals and patients focusing on the impact of age, genes and training intensity. A further step in this research will be to investigate the impact of age, genes, training intensity and history of tick-bourne disease on endurance performance in elite endurance athletes. We are planning a project with a two-step model. In step one we will, in a cross-sectional study design, investigate potential relationships between age, training intensity, training volume, genes, exosomes and history of tick-bourne disease and physiological variables and endurance performance. In step two we will investigate differences in training adaptation by observing and monitoring all training done by the participants during a 6-months period. The participants will be tested for several physiological variables before, after 3- months and after this period. We will also investigate the impact of age, training intensity, training volume, genes and history of tick-bourne disease on the results from the physiological tests and performance.

DETAILED DESCRIPTION:
The study will be designed in a two-step model. In the first step, we will investigate potential relationships between age, genes, exosomes, miRNA, training intensity, and history of tick-borne disease, and physiological laboratory-tests and performance in a roller-skiing performance test. This study will have a cross-sectional design. In the second step we will examine potential differences in training adaptations to a 6-months observation of self-selected training. We then will categorize the athletes into three groups, based on training volume and training intensity. We will then investigate possible relationships between training volume and training intensity and physiological variables, genes, age and possible history of tick-bourne disease.

STEP 1: Cross-sectional study:

Since the aim of the study is to investigate effects of age, genes, exosomes, training and history of tick-borne disease on training adaptations and endurance performance in elite endurance athletes, we will recruit active cross-country skiers from 16 - 50 years. These athletes have shown to have some of the highest aerobic capacities in the world (Ingjer, 1991).

Both males and females will be included for participation in this project, and we will try to include equal amount of both sexes. The athletes will be recruited from relevant, cross-country skiing milieus in Southeast Norway by open invitation and advertisement. Invited athletes must sign a declaration for participation and a declaration of health status, before participation. In the declaration for participation, the athletes will be informed briefly about the background of this project, which tests they are going to take, and how these tests will be performed and how the results are being contained and presented.

Statistical analysis will be as descriptive statistics, and simple and multiple regressions- and correlation analysis in the cross-sectional study.

STEP 2: 6-months training observation:

Recruitment routines, inclusion- and exclusion criteria will be the same as in STEP 1.

The athletes will first undergo a week of testing and registration (like STEP 1) at the end of the competitive season. During the 6-months period, the athletes will register all normal training in training diaries, and most importantly by use of heart rate measures. The researchers will not assign the participants to a certain training program or intervention, but just observe and register their training already planned out by themselves and/or their trainer(s). We will then examine the effects of this training on physiological variables and cross-country skiing performance

The first tests will include the following:

* physiological determinants as described in Støren et al. (2012; 2013; 2014) and Sunde et al. (in progress)
* blood samples for the analyze of genes, types of exosomes and its cargo, miRNA and history of tick-borne disease The same tests will be used after 3 months into the training period, and post observation. Tests and test procedures will be specified later.

Statistical analysis will be as descriptive statistics, hypothesis testing as General Linear Models ANOVA (repeated measurements), and simple- and multiple regressions- and correlation analysis to examine increase or decrease in relation to age, gender, physical capacity and genes.

Tests and test procedures:

The same test procedures will be followed in both STEP 1 and STEP 2 of the project, and pre-, mid- and post-test. All tests will be executed in two following days.

Day 1:

* Registration of body weight, body height and BMI, and blood samples for exosomes, genes and tick-borne disease
* Maximal jump tests (SJ, CMJ and CMJas)
* VO2max test in running, followed by blood samples for exosomes
* Performance field-test in roller skiing

Day 2:

* LT-test and energy cost of double poling (Cp)
* VO2peak in double poling
* Blood samples for exosomes
* 1RM half-squat, followed by blood samples for exosomes
* 1RM pull down

DAY 1:

When the athletes arrives, body weight and body height will be measured. Blood samples will be taken for analysis of exosomes, genes and tick-borne disease.

Blood samples and genetic analysis To examine the effects of exosomes, genes and history of tick-borne disease on training adaptation and endurance performance among elite endurance athletes, it will be necessary to gather blood samples for examination of genetic variation, exosome cargo, exosome content and antibodies for tick-borne diseases.

The field, Exercise Genomics, explore the variation in single candidate genes relation to physiological responses to exercise in a population. Therefore, it is relevant to apply research on genes relation to training adaptations and human endurance performance, but also in relation to health-related physical activity. We also want to analyze volume and types of exosomes in response to training, with a focus on content of miRNA, proteins and/or DNA as biological markers for physiological training response.

In this research project we need blood samples from recruited cross-country skiers to examine genetic variations, which have been related to cause an effect on physiological responses like fat oxidation, glucose utilization, insulin sensitivity, muscle hypertrophy, VO2max and blood pressure. The exosomes will be isolated from plasma by an ultracentrifugation method.

Blood samples for analysis of biological markers We want blood samples (EDTA-blood) from all participants. Blood samples will be taken in relation to the training interventions, and will be used for DNA isolation, DNA analysis, exosome isolation from plasma and isolation of antibodies from plasma.

Jumping variables (SJ, CMJ, CMJas):

After arrival and registration of body weight and body height, the athletes will be instructed to perform a 10-minutes self-conducted warm-up before testing. For measuring jump height, we will use a force plate and the Muscle Lab v.2 system (Ergotest Technology, Langesund, Norway) The first jump procedure will be by measuring squat jump (SJ) height. The subjects' starts with a 90° knee angle, with a forward leaned position and with their hands attached to the hips. The subjects' will then jump with maximal force, without any counter movement in the knees or hips. The subjects perform minimum three and maximum six jump with maximal force, where the highest jump will be registered as the result.

After this, the subjects will perform the second jumping procedure, who will be the counter-movement jump (CMJ). The athletes start in an upright position with their hands attached to the hips. They will thereafter perform a maximal jump with plyometric movement. The subjects perform minimum three and maximum six jump with maximal force, where the highest jump will be registered as the result.

The last jump procedure is the counter movement jump with arm movement. The subjects starts in the position like CMJ, but are now allowed to use the arms. They will be instructed to perform a jump with maximal force. The subjects perform minimum three and maximum six jump with maximal force, where the highest jump will be registered as the result.

The subjects' are given three minutes rest between each jumping procedure.

VO2max in running:

The test will be performed on a motorized Woodway PPS55-treadmill (Waukesha, WI, USA), calibrated for elevation and speed. A Cortex MetaLyzer II (Cortex Biophysik GmbH, Leipzig, Germany) measures VO2 every 10 s through the test. The subjects' will be instructed to perform a 10-minutes self-conducted warm-up before testing.

The test starts at 8 - 12 km/h, and a 6% elevation. A 1% elevation increase will be performed up to 8%. From there, only speed increases with 0,5 km/h every 30 second until voluntary exhaustion.

Contra indications during testing will end the test. The participants are allowed to stop the test at any given time.

To evaluate if VO2max is reached, we will use the following criteria: flattening of the O2-curve, RER > 1.05, 3 - 5 beats under the athlete's maximal heart rate (HRmax), Borg scale > 16 and blood lactate levels > 8.0 mmol/l.

Time-trial performance test on roller skies The participants will be instructed to perform a minimum 15 minutes self-conducted warm-up before test. They will use their own roller-skiing equipment during this test. Before testing, the athletes will be informed to use Swenor 2-wheels, or equal, during this test to prevent any differences in rolling resistance.

During this test, the athletes participate in randomly assigned pairs, with a 1-minute start interval between subjects. They will perform six laps of 940 meters, as fast as they can, using only the double-poling technique. No drafting is allowed. Stopwatches register performance time.

The total time used in this time-trial will be used as result from this test. Heart rate will be monitored by the athletes private watches, and registered immediately after finish.

DAY 2:

Lactate threshold (LT) og cost of poling (Cp) during double-poling The test will be performed on a Rodby RL2500E - treadmill with rubber belts (Rodby Innovation, Vänge, Sweden), special made for double poling. The participants will perform a minimum 10 minutes self-conducted warm-up before testing, and for familiarization to the treadmill.

Lactate, VO2 and RER will be measured during several 4-minute submaximal work periods (minimum 3 and maximum 6) at 4% inclination. All the athletes will use the same roller-skies, but they will use their own poles and shoes during the test. The procedure for this test will be as follows:

* Work period 1: The workload will represent approximately 60% HRmax. The speed of the treadmill will be set to 11.5 km/h and 6 - 7 km/h for males and females respectively, and will be held constant through the 4-minute work period. After 4 minutes, the treadmill stops and lactate measuring will be proceeded.
* Work period 2, 3 and 4 (eventually 5 and 6): The speed will increase progressively (evaluated by research-personal) through the work periods, until blood lactate exceeds estimated LT-values (LT = warm-up lactate value (taken after the first work period) + 2,3 mmol/l).
* HR and VO2 will be measured every 20 second from the 3.00 minute point in every work period (3.00 / 3.20 / 3.40).

Blood lactate is measured by a Lactate Scout+ apparatus (Senslab, EKF Diagnostics, Germany), which is based on whole blood analysis.

Contra indications during testing will end the test. The participants are allowed to stop the test at any given time.

Registration of VO2 during the work periods are later used for calculations of Cp at 70% Vo2max.

VO2peak double poling The test will be performed at least 5 minutes after the LT-test on the same treadmill specialized for double poling. All the athletes will use the same roller-skies, but they will use their own poles and shoes during the test. VO2, HR and RER will be measured continuously during this test.

The test will proceed as follows:

* The speed is set to 7 km/h for both males and females, at a 6 % inclination and is held constant through the whole test.
* The speed progressively increase by 1 km/h every minute for males and females, until exhaustion.

The three continuously highest VO2 measures will be used for calculation of VO2max. The test will be followed by registration of blood lactate (as described earlier), Borg scale, RERpeak and HRpeak.

1RM half squat:

For this test, a Precor smith-machine (Precore, Woodinville, WA, USA) will be used. The athletes will be given at least 60 minutes rest between last test, and this test. The participants will follow a standardized warm-up procedure as follows:

* 10 repetions à 50% 1RM,
* 5 repetions à 60% av 1RM,
* 3 repetions à 70% av 1RM
* 2 repetions à 80% av 1RM. A 3-minute rest period will be given between every work period. The participants will be instructed to lift with maximal speed from the first workload, for measuring muscle power. MuscleLab v. 2 (Ergotest Technology, Langesund, Norway) will measure power during the test.

After the standardized warm-up, the workload will increase progressively until 1RM is reached. In this part of the test, the participants only perform one repetion pr. workload.

1RM pull down: A Gym2000 pull-down machine (Gym2000 AS, Vikersund, Norway) will be used for this test. The protocol for this test is identical to the 1RM half-squat protocol.

ELIGIBILITY:
Inclusion Criteria:

* age between 16 and 50
* active competition athletes competing on a national level or above
* athletes who write training diaries

Exclusion Criteria:

* Sickness and/or injury who contra indicates normal training and maximal testing.
* An on-going infection or injury.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cross-country skiers at high national or international level
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Time trail cross-country roller skiing performance | Change from baseline performance at 3-months and at 6-months
  Testing of seconds used in a predefined track
Maximal oxygen consumption | Change from baseline maximal oxygen uptake at 3-months and at 6-months
  Standard ergospirometrical incremental test in running and double-poling

SECONDARY OUTCOMES:
Lactate threshold in double poling | Change from baseline lactate threshold at 3-months and at 6-months
  Onset of blood lactate accumulation in an incremental interval protocol
Double poling economy | Change from baseline economy at 3-months and at 6-months
  Ergospirometrical measurement of oxygen consumption per meter poling
Maximal strength | Change from baseline maximal strength at 3-months and at 6-months
  Kilograms measured in one repetition maximum in half-squat and pull-down
Jump height | Change from baseline jump height at 3-months and at 6-months
  Centimeters measured on force platform in squat jump, counter movement jump and countermovement jump with armswing
Genotypes | Baseline
  Distribution of alleles for candidate genes derrived from blood samples
Tick-bourne disease | Baseline
  Blood markers for previous tick-bourne disease
Exosomes | Baseline
  Quantifying number of exosomes in blood immediately before and after maximal aerobic work and maximal strength tests
Training volume | Change from baseline training volume at 3-months and at 6-months
  Registration of training volume in hours from training diaries
Training intensity | Change from baseline training intensity at 3-months and at 6-months
  Registration of training intensity by use of heart rate measures corresponding to the training intensity scale made by the Norwegian Olympic Sports Center.
Age | Baseline
  Age in years
Maximal power | Change from baseline power at 3-months and at 6-months
  Maximal power in watt in half-squat and pull-down

CONTACTS AND LOCATIONS:
Overall Officials: Pål Augestad, PhD, Study Chair — University of South-Eastern Norway
Locations (1):
- Telemark University College, Bø, Telemark, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Storen O, Bratland-Sanda S, Haave M, Helgerud J. Improved VO2max and time trial performance with more high aerobic intensity interval training and reduced training volume: a case study on an elite national cyclist. J Strength Cond Res. 2012 Oct;26(10):2705-11. doi: 10.1519/JSC.0b013e318241deec. PMID 22124353
- [Background] Ingjer, F. Maximal oxygen uptake as a predictor of performance ability in women and men elite cross-country skiers. Scand. J. Med. Sci. Sports. 1: 25-30, 1991.
- [Background] Storen O, Ulevag K, Larsen MH, Stoa EM, Helgerud J. Physiological determinants of the cycling time trial. J Strength Cond Res. 2013 Sep;27(9):2366-73. doi: 10.1519/JSC.0b013e31827f5427. PMID 23238091
- [Background] Storen O, Ronnestad BR, Sunde A, Hansen J, Ellefsen S, Helgerud J. A time-saving method to assess power output at lactate threshold in well-trained and elite cyclists. J Strength Cond Res. 2014 Mar;28(3):622-9. doi: 10.1519/JSC.0b013e3182a73e70. PMID 23942166